CLINICAL TRIAL: NCT00048776
Title: Safety and Efficacy of Pletal (Cilostazol) for the Treatment of Juvenile Primary and Secondary Raynaud's Phenomenon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-01-336
Record Dates: First submitted 2002-11-07; First posted 2002-11-11 (Estimated); Last update posted 2005-07-19 (Estimated); Status verified 2005-07

CONDITIONS: Raynaud's Disease
Keywords: Secondary Raynaud's; circulatory; vascular; scleroderma; lupus; mixed connective tissue disease
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Diffuse; Mixed Connective Tissue Disease | interventions — Cilostazol

INTERVENTIONS:
Drug: Pletal

SUMMARY:
Juvenile secondary Raynaud's (ray-knows) Phenomenon is a disorder of the blood vessels in the fingers and sometimes can affect the toes, nose, or ears. Children with secondary Raynaud's Phenomenon have an underlying condition such as systemic lupus, scleroderma, or mixed connective tissue disease. When children with secondary Raynaud's are exposed to chilly or cold conditions from weather, cold temperatures, or even holding cold items from the refrigerator, their fingers may become cold, numb, hurt, and/or turn purple or white. The investigational drug, Pletal(cilostazol), which has been approved for other conditions, inhibits the ability of one type of blood cell, platelets, to form blood clots, and also widens narrowed blood vessels. It has been used in a variety of other conditions in which blood flow is decreased. This study will test the safety and effectiveness Pletal(cilostazol) to lessen the severity of the symptoms and decrease the number of secondary Raynaud's episodes in juvenile patients.

ELIGIBILITY:
Inclusion Criteria

* 5 to 16 years old
* fulfill diagnostic criteria for primary or secondary Raynaud's

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75
Dates: Start 2001-10; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Advanced Medical Clinical Therapeutics, Anchorage, Alaska
  - Advanced Medical Research Institute, Fresno, California
  - Madera Family Medical Group, Madera, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - LaRabida Children's Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Children's Hospital, Omaha, Nebraska
  - Asthma & Allergy Research Center, Newark, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Children's Hospital of Buffalo, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - New York Medical College, Valhalla, New York
  - Jobst Vascular Center, Toledo, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Monarch Research Associates, Norfolk, Virginia
  - Children's Hospital and Regional Medical Center, Seattle, Washington